CLINICAL TRIAL: NCT03948867
Title: Stroke Prevention With Hydroxyurea Enabled Through Research and Education (SPHERE): A Prospective Trial to Reduce Primary Stroke in Children With Sickle Cell Anaemia
Brief Title: Stroke Prevention With Hydroxyurea Enabled Through Research and Education (SPHERE)
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: Bugando Medical Centre (Unknown); The American Society of Hematology (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SPHERE
Record Dates: First submitted 2019-02-08; First posted 2019-05-14 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Sickle Cell Anemia in Children
Keywords: Sickle Celll Anemia; Transcranial Doppler; Tanzania; Hydroxyurea; Stroke
MeSH Terms: conditions — Stroke | interventions — Hydroxyurea

STUDY DESIGN:
Intervention Model Description: The cohort will be divided into two arms based on the initial screening TCD result: 1) those who have a normal initial screening TCD and will be an observation/control cohort; and 2) those who have an elevated initial screening TCD (either conditional or abnormal TAMV) and will be a treatment cohort that receives open-label hydroxyurea therapy as per the dosing and administration schedule
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Elevated Initial Screening TCD (Experimental): Those who have an elevated initial screening TCD (either conditional or abnormal TAMV) and will be a treatment cohort that receives open-label hydroxyurea therapy as per the dosing and administration schedule.
  Interventions: Drug: Hydroxyurea; Diagnostic Test: Elevated Arm TCD Examination
- Normal Initial Screening TCD (Experimental): Those who are found to have a normal TCD at enrolment are a part of the observation/control cohort and will undergo repeat TCD every 12 months after enrolment. If the TCD at 12 months has changed to an elevated velocity (conditional or abnormal), the study participant will be reassigned to the elevated initial screening TCD arm and can begin study treatment (hydroxyurea), but will not be included in the primary endpoint analysis.
  Interventions: Diagnostic Test: Normal Arm TCD Examination

INTERVENTIONS:
Drug: Hydroxyurea — Hydroxyurea treatment will be provided to reduce stroke risk. Hydroxyurea treatment will be started at a fixed dose of 20.0 ± 5.0 mg/kg/day, followed by escalation to maximum tolerated dose (MTD).
  Arms: Elevated Initial Screening TCD
Diagnostic Test: Elevated Arm TCD Examination — TCD examination on children with SCA between ages 2 and 16 years of age will be completed to evaluate their risk of stroke.
  For children with elevated velocities at initial screening or at 1 Year who receive hydroxyurea therapy, TCD examinations will occur every 6 ± 2 months.
  Arms: Elevated Initial Screening TCD
Diagnostic Test: Normal Arm TCD Examination — TCD examination on children with SCA between ages 2 and 16 years of age will be completed to evaluate their risk of stroke. TCD examination for all participants will occur at initial screening, at Year 1 (12 ± 3 months), and Year 2 (24 ± 3 months). Children with normal TCD velocities at initial screening will undergo repeat TCD 12 months after enrolment. If the TCD at 12 months has changed to an elevated velocity (conditional or abnormal), the child can begin study treatment (Hydroxyurea).
  Arms: Normal Initial Screening TCD

SUMMARY:
This study will 1) Evaluate the prevalence of elevated (conditional or abnormal) transcranial Doppler (TCD) velocities in a cross-sectional analysis of children with Sickle Cell Anemia (SCA) living in Tanzania; 2) Obtain longitudinal data on TCD velocities in this population; and 3) Measure the effects of hydroxyurea therapy on TCD velocities and associated primary stroke risk.

DETAILED DESCRIPTION:
Stroke Prevention with Hydroxyurea Enabled through Research and Education (SPHERE) is a single-center prospective phase 2 pilot study. It will enroll a convenience sample of children with SCA, obtain cross-sectional baseline data at enrolment, and follow them as a prospective cohort for a period of 24 months. The cohort will be divided into two arms based on the initial screening TCD result: 1) those who have a normal (less than 170 cm/sec time averaged mean velocity (TAMV)) initial screening TCD and will be an observation/control cohort; and 2) those who have an elevated initial screening TCD (either conditional (170-199 cm/sec) or abnormal (greater than or equal to 200 cm/sec) TAMV) and will be a treatment cohort that receives open-label hydroxyurea therapy as per the dosing and administration schedule. Those who are found to have a normal TCD at enrolment and are part of the observation/control cohort will undergo repeat TCD 12 months after enrolment. If the TCD at 12 months has changed to an elevated velocity (conditional or abnormal), the study participant can begin study treatment, but will not be included in the primary endpoint analysis. The primary hypothesis is after 12 months of hydroxyurea therapy, children with conditional TCD velocities will achieve a mean decrease of >15cm/sec from their baseline TCD TAMV.

ELIGIBILITY:
Inclusion Criteria:

* Willingness to sign informed consent
* Willingness to follow all study procedures
* Available for study visits for the duration of the study and no plans to move away from study center.
* Confirmed diagnosis of Sickle Cell Anemia (SCA) by haemoglobin electrophoresis.
* Able to take oral medication and follow hydroxyurea treatment schedule.

Exclusion Criteria:

There are no permanent exclusion criteria for participants to enroll in the screening TCD portion of SPHERE. Temporary, time-limited exclusion criteria for the screening TCD portion include the following:

* Febrile illness within the past two weeks. (Temporary Exclusion)
* Hospitalized within the past two weeks. (Temporary Exclusion)
* Transfusion within the past two weeks. (Temporary Exclusion)

Patients who enroll in the screening portion, have a conditional or abnormal TCD, and are eligible to start hydroxyurea will be excluded from receiving study treatment if they meet any of the following criteria:

* Abnormal pre-enrolment laboratory values (Temporary Exclusion)
* Known medical condition making participation ill-advised.
* Known allergic reactions to components of hydroxyurea.
* Previous history of stroke.
* Currently pregnant or lactating.

Ages: 2 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 202 (Estimated)
Dates: Start 2019-04-24 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Prevalence of Elevated TCD | Baseline
  Determine the prevalence of elevated (conditional or abnormal) transcranial Doppler (TCD) velocities in a cross-sectional analysis of children with Sickle Cell Anemia (SCA) living in Tanzania
Change in Primary Stroke Risk | Up to 12 Months at Month 12
  Transcranial Doppler ultrasound (TCD) will be used to measure the change in the TAMV of arterial blood flow in the 4 major intracranial arteries bilaterally from study enrollment to 12 months after study enrollment.

SECONDARY OUTCOMES:
Laboratory and Clinical Correlates | Up to 24 Months
  Identify laboratory and clinical correlates of elevated TCD velocities such as age, haemoglobin concentration, foetal haemoglobin, oxygen saturation, splenomegaly, history of acute chest syndrome, and previous malaria infection
Change in Hemoglobin Concentration | 6 Months
  For those receiving hydroxyurea, the change in hemoglobin between baseline hemoglobin and follow up hemoglobin when a participant has reached maximum tolerated dose of hydroxyurea.
Effect of Splenomegaly and Malaria Infections | Up to 24 Months
  Incidence of splenomegaly and malaria infection with rapid or laboratory malaria testing will be performed for any child presenting with fever. Incidence will be reported in the number of cases per 100 patient years. Abdominal ultrasound with splenic volume will be performed annually for all study participants. Quantify the degree of hypersplenism or autoinfarction and any association with malaria complications of SCA will be analyzed.
Prevalence of Co-inherited G6PD and Alpha Thalassemia | One time at Baseline
  DNA will be collected at baseline to determine the prevalence of co-inherited hematologic diseases such as G6PD and alpha thalassemia.
Hydroxyurea Area Under the Curve (AUC) | One time at 24 Months (Study Exit)
  For those receiving hydroxyurea, the AUC will be assessed after the patient has reached MTD.
Single Nucleotide Polymorphisms Associated with Change in Percent Hemoglobin F on Hydroxyurea | One Time at 24 Months (Study Exit)
  For those receiving hydroxyurea, we will identify single nucleotide polymorphisms that are associated with a greater change in hemoglobin F percent in response to hydroyxurea therapy.

CONTACTS AND LOCATIONS:
Locations (2):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States
- Bugando Medical Centre, Mwanza, Tanzania

REFERENCES:
- [Derived] Ambrose EE, Latham TS, Songoro P, Charles M, Lane AC, Stuber SE, Makubi AN, Ware RE, Smart LR. Hydroxyurea with dose escalation for primary stroke risk reduction in children with sickle cell anaemia in Tanzania (SPHERE): an open-label, phase 2 trial. Lancet Haematol. 2023 Apr;10(4):e261-e271. doi: 10.1016/S2352-3026(22)00405-7. Epub 2023 Mar 1. PMID 36870358